CLINICAL TRIAL: NCT07283601
Title: Mindfulness-Based Stress Reduction for Disaster-Affected Women: A Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial of Mindfulness-Based Stress Reduction for Reducing Perceived Stress in Women Impacted by Large-Scale Disasters
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Leyla SEZGİN, Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: Disaster; Muş Alparslan Universty (Other: Muş Alparslan Universty)
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Mindfulness, Woman, Stress, Disaster
Keywords: mindfulness, woman, stress, disaster

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the experimental group will receive an 8-week Mindfulness-Based Stress Reduction (MBSR) program designed to reduce perceived stress and enhance emotional resilience.
  The intervention will consist of:
  Weekly group sessions (2-2.5 hours each) led by a certified MBSR instructor,
  Daily home practice (30-45 minutes per day), supported by guided meditation recordings.
  Each session will include:
  Mindfulness meditation focused on present-moment awareness,
  Body scan exercises to enhance bodily awareness,
  Gentle yoga and stretching,
  Breathing and relaxation techniques, and
  Group discussions and reflection to integrate mindfulness into daily life.
  Participants will be encouraged to maintain a daily mindfulness routine and record their practice in provided logs.
  Interventions: Behavioral: MBSRP
- Control (No Intervention): Participants assigned to the control group will not receive any intervention during the study period.
  They will complete the same assessment measures as the experimental group at baseline, post-intervention (week 8), and follow-up (if applicable).
  This group serves as a comparison to evaluate whether changes in perceived stress are specifically attributable to the Mindfulness-Based Stress Reduction (MBSR) program rather than natural recovery or time effects.
  After the completion of data collection, participants in the control group will be offered the opportunity to participate in the MBSR program (wait-list control condition) for ethical considerations.

INTERVENTIONS:
Behavioral: MBSRP — The intervention consists of an 8-week Mindfulness-Based Stress Reduction (MBSR) program designed to reduce perceived stress and promote emotional resilience among disaster-affected women.
  Each session will last approximately 2 to 2.5 hours per week, conducted by a certified MBSR instructor in small groups of 10-15 participants.
  The program includes:
  Mindfulness meditation,
  Body scan exercises,
  Gentle yoga and stretching,
  Breathing awareness and relaxation techniques, and
  Group discussions and reflections to integrate mindfulness practices into daily life.
  Participants will be asked to complete 30-45 minutes of daily home practice using guided meditation recordings.
  The primary goal of the intervention is to decrease perceived stress and enhance psychological well-being among women who have experienced large-scale disasters.
  Arms: Intervention

SUMMARY:
Hypothesis:

Women affected by large-scale disasters who participate in an eight-week Mindfulness-Based Stress Reduction (MBSR) program will experience significantly lower perceived stress levels compared to those in the control group without intervention.

DETAILED DESCRIPTION:
Objective: This study aims to describe the effect of the Mindfulness-Based Stress Reduction Program (MBSRP) administered in relation to post-disaster stress.

Material and Method: The present study was carried out by using a quasi-experimental design with 35 participants in the intervention group and 33 in the control group. Personal Information Form, Mindful Attention Awareness Scale (MAAS), and Perceived Stress Scale (PSS) were employed in the data collection process. The women in the intervention group underwent an 8-week Mindfulness Stress Reduction Program. Data were collected through pretests and posttests.

Descriptive statistics were used for data analysis. Independent samples t-test and dependent samples t-test were utilized for the control and intervention groups. The relationship between continuous variables was analyzed by using Pearson Correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged 18-65 years. Have been directly affected by a large-scale disaster (e.g., earthquake, flood, fire, or similar event) within the past 12-24 months.

Report moderate or high perceived stress levels (Perceived Stress Scale [PSS-10] score ≥ 14).

Able to attend weekly MBSR sessions for 8 consecutive weeks. Willing to provide written informed consent to participate in the study.

Exclusion Criteria:

Current diagnosis of severe psychiatric disorder (e.g., psychosis, bipolar disorder, severe major depression).

Ongoing psychotherapy or psychopharmacological treatment for stress, anxiety, or depression at the time of enrollment.

Prior participation in any mindfulness or meditation-based program within the last 6 months.

Presence of a serious medical condition (e.g., uncontrolled hypertension, cardiovascular disease) that could interfere with participation.

Pregnancy or postpartum period (<6 months), if it affects stress levels or participation.

Inability to understand study instructions or complete questionnaires in Turkish.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — WOMEN
Enrollment: 70 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure: Change in perceived stress level measured by the Perceived Stress Scale (PSS-10) from baseline to week 8 | Baseline (Week 0) - before the start of the intervention Post-intervention (Week 8) - immediately after completion of the 8-week MBSR program Follow-up (Week 12 or Week 16) - four to eight weeks after the intervention to assess maintenance of effects
  Primary Outcome Title:
  Perceived Stress Level
  Description:
  The primary outcome will be the change in perceived stress levels from baseline to 8 weeks after the intervention.
  Measurement Tool:
  Perceived Stress Scale (PSS-10), a validated 10-item self-report questionnaire that measures the degree to which situations in one's life are appraised as stressful.
  Time Frame:
  Baseline (Week 0) and Post-intervention (Week 8)
  Scoring and Interpretation:
  Total scores range from 0 to 40, with higher scores indicating greater perceived stress. A decrease in the mean PSS-10 score from baseline to week 8 in the intervention group compared to the control group will indicate a positive treatment effect.
  Type of Outcome:
  Continuous variable (mean score difference between groups)

CONTACTS AND LOCATIONS:
Locations (1):
- Muş Alparslan University, Merkez, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD Sharing Plan Description:
  De-identified individual participant data (IPD) that underlie the results reported in this study will be shared upon reasonable request after publication of the main findings. The shared data will include demographic variables, baseline characteristics, outcome measures (e.g., Perceived Stress Scale scores), and intervention adherence information.
  Data will be available to qualified researchers for secondary analyses that are consistent with the original study objectives. Requests for access must include a methodologically sound proposal and ethical approval.
  Data will be shared through a secure data repository or institutional data-sharing agreement, ensuring participant confidentiality according to relevant data protection regulations (e.g., GDPR, national ethics standards).
  Time Frame for Data Sharing:
  Beginning 6 months after publication of the primary results and available for up to 3 years following that date.